CLINICAL TRIAL: NCT07127068
Title: Investigation of the Effects of Omega-3 Supplementation in Chronic Kidney Disease Patients Diagnosed With Coronary Artery Disease and Dyslipidemia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Eda BALCI, Lecturer, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDABALCI2025
Record Dates: First submitted 2025-08-04; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-02

CONDITIONS: Omega 3 Fatty Acids; Coronary Arterial Disease (CAD); Chronic Kidney Disease(CKD)
Keywords: chronic kidney disease; omega 3 fatty acids; coronary arterial disease; dyslipidemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients taking omega 3 fatty acids (Experimental): This group will be asked to use 2 capsules containing 2000 mg (720 mg EPA, 480 mg DHA) omega 3 daily for 12 weeks. The total of these capsules taken in the morning and evening provides the daily dose.
  Interventions: Dietary Supplement: Omega-3 Suplementation
- Control (Experimental): This group will be the control group. No supplements will be used in this group. Only the appropriate diet list will be applied.
  Interventions: Other: No intervention

INTERVENTIONS:
Dietary Supplement: Omega-3 Suplementation — The intervention group will receive a daily oral supplementation of 2000 mg omega-3, which will not be administered to the control group. Blood samples will be collected from all participants at baseline and at the end of the study to evaluate selected serum parameters. To minimize nutritional variability, individualized diets appropriate for coronary artery disease and chronic kidney disease were prescribed to both groups at the beginning of the study. Unlike many other intervention studies, this trial specifically targets end-stage renal disease patients and includes an evaluation of the intervention's impact in relation to dialysis initiation.
  Arms: Patients taking omega 3 fatty acids
Other: No intervention — Participants in the control group will not receive any dietary supplementation. Blood samples will be collected at baseline and at the end of the study to assess selected biochemical parameters. Standard dietary care appropriate for coronary artery disease and chronic kidney disease will be maintained throughout the study.
  Arms: Control

SUMMARY:
Chronic kidney disease (CKD) is characterized by the slow, progressive, and irreversible loss of kidney function. Uremic toxins in CKD patients trigger an inflammatory response driven by various cytokines, chemokines, and other inflammatory molecules. As a result, increased oxidative stress and tissue damage are observed. In such an inflammatory environment, CKD patients are at higher risk of mortality due to the occurrence of adverse cardiovascular events. Omega-3 fatty acids are long-chain polyunsaturated fatty acids such as α-linolenic acid (ALA, 18:3), eicosapentaenoic acid (EPA, 20:5), and docosahexaenoic acid (DHA, 22:6). Omega-3 fatty acids are essential fatty acids because they cannot be synthesized in the body. There is increasing evidence that omega-3 fatty acids play a role in regulating inflammation and immune response by reducing the production of monocyte proinflammatory cytokines interleukin-1 (IL-1), IL-6, and TNF-α. Omega-3 has also been shown to alter abnormal lipid metabolism, reduce platelet aggregation, improve homocysteine levels, and improve endothelial function, blood pressure, heart rate, and oxidative stress.

This study, which aims to observe the effectiveness of omega-3 supplementation in individuals who must have a diet low in omega-3 fatty acids due to certain dietary restrictions (especially fish), will be conducted at the Health Sciences University Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Education Research Hospital. 60 patients between the ages of 50-75 with chronic kidney disease diagnosed with coronary artery disease and dyslipidemia will be included in the study. The study will include patients with stage 2-4 chronic kidney disease who have a history of dyslipidemia and coronary artery disease, a glomerular filtration rate (GFR) of 20-60 ml/min, a body mass index (BMI) of 18-30 kg/m2, are 50-75 years old, and have LDL cholesterol >70 mg/dl despite using equal doses of statins for at least 3 months. Ethics committee approval for the study was obtained from the Istanbul Medipol University "Non-Interventional Clinical Research" ethics committee. Randomly selected participants of similar sizes will be randomly divided into 2 groups. Group A (intervention group) will be asked to use 2 capsules containing 2000 mg (720 mg EPA, 480 mg DHA) omega 3 daily for 12 weeks. The total of these capsules taken in the morning and evening will provide the daily dose. Group B will be the control group. No supplement will be used in this group. Clinical, biochemical and functional status data of each participant will be obtained at the beginning of the study and after the 12-week intervention. Apart from the parameters checked in routine tests (Total cholesterol (mg/dL), LDL-C (mg/dL), HDL-C (mg/dL), triglyceride (mg/dL), CRP (mg/L), fasting blood glucose (mg/dL), calcium (mg/dL), phosphorus (mg/dL), sodium (mg/dL), potassium (mg/dL), Creatine, Urea, Uric acid), Homocysteine, IL-6, TNF-a, Superoxide dismutase (SOD) and Malondialdehyde (MDA) levels will be analyzed in Istanbul Beykent University Multidisciplinary Laboratory. Anthropometric measurements (height, weight) of the patients will be taken. In addition, the food consumption records and food consumption frequencies of the patients will be evaluated with the BeBIS program.

DETAILED DESCRIPTION:
Chronic kidney disease is defined as the detection of kidney damage markers in urine, blood and radiological examinations, regardless of the glomerular filtration rate, or the glomerular filtration rate (GFR) being below 60 ml/min/1.73 m² and the continuation of the relevant findings for at least 3 months. CKD leads to certain clinical outcomes by the body's inability to perform its metabolic and endocrine functions, the inability to regulate fluid-electrolyte balance, and affecting almost every system in the body. Metabolic abnormalities including hyperphosphatemia, secondary hyperparathyroidism, hypocalcemia and dyslipidemia are seen in advanced CKD patients. Together with chronic inflammation, increased oxidative stress and malnutrition associated with CKD, these abnormalities increase cardiovascular risk. As the glomerular filtration rate (GFR) decreases and kidney disease progresses from GFR category G1 to G5, the proportion of CKD patients who die from cardiovascular disease increases. Omega-3 fatty acids are in the polyunsaturated fatty acid class. There are three omega-3 fatty acids that are important in human physiology and nutrition; These are α-linolenic acid (ALA; 18:3), EPA (20:5) and DHA (22:6) (Bowen et al., 2016). While ALA is found in vegetable oils such as flaxseed, canola, olive oil and walnuts, EPA and DHA are especially abundant in oily fish such as tuna, salmon and trout. Omega-3 fatty acids are essential fatty acids because they cannot be synthesized in the body. CKD is a chronic inflammatory process. Serum proinflammatory protein levels are 10 times higher in these patients than in the normal population. It is known that CRP levels are higher in both predialysis patients and patients on dialysis compared to the normal population. Increased serum proinflammatory protein levels have many systemic effects such as fever, loss of appetite, nausea, vomiting, increased atherosclerotic plaque development and blockade of albumin synthesis. It is known that especially CRP, tumor necrosis factor alpha (TNF-α), Interleukin (IL)-1 and IL-6 levels are high in these patients. These high pro-inflammatory protein levels cause malnutrition and atherosclerosis in patients, paving the way for mortality and morbidity. Omega-3 has properties related to the inhibition of inflammation and is thought to be effective in patients with chronic kidney disease. EPA and DHA are the precursors of molecules responsible for the suppression of the inflammatory process, as well as improving abnormal lipid metabolism, reducing platelet aggregation, improving endothelial function, blood pressure, heart rate and oxidative stress.

The aim of the study is to investigate the effectiveness of omega-3 supplementation on serum lipid levels, homocysteine, inflammatory and oxidative stress biomarkers in chronic kidney disease patients whose consumption of omega-3 rich foods is limited due to dietary restrictions and whose blood lipids do not reach the desired level despite using antilipidemic drugs. In patients with stage 2-4 chronic kidney disease, fish consumption, which is the food that contains the most omega-3, is very limited. Because these patients' serum phosphorus levels and protein intake are limited in their diet programs in order to be at the desired level. At the same time, other foods rich in omega-3 are restricted in terms of potassium content (e.g. walnuts). Therefore, the serum omega-3 levels of the patients are also low. Our aim is to investigate the effects of omega-3 supplementation in this patient group. According to the results of the study, adding omega-3 supplementation to the patients' treatments may yield positive results in terms of disease progression.

This study will be conducted at the Health Sciences University Dr. Siyami Ersek Thoracic Cardiovascular Surgery Training and Research Hospital. 60 patients with chronic kidney disease diagnosed with coronary artery disease and dyslipidemia, aged between 50-75 years, will be included in the study.

Inclusion Criteria; Diagnosed with dyslipidemia Diagnosed with type 2 diabetes Having a history of coronary artery disease Glomerular filtration rate 20-60 ml/min Stage 2-4 chronic kidney disease patients Body Mass Index (BMI) 18-30 kg/m2 Age between 50-75 Patients with LDL cholesterol >70 mg/dl despite using equal doses of statin group drugs for at least 3 months (desired value for these patients according to the European Association of Cardiology) Exclusion Criteria Having active inflammatory disease Having chronic inflammation such as active hepatitis, human immunodeficiency virus (HIV)(+) using anti-inflammatory drugs Having liver disease - increased liver enzymes Receiving dialysis treatment Those planned for transplantation Those using fish oil and other antioxidant drugs in the last 3 months Pregnant and breastfeeding women Those with neurological and psychiatric diseases More than 1 serving per week Individuals who consume foods high in omega 3 fatty acids such as fish and walnuts Patients with a high risk of bleeding (Those using Bivalirudin group drugs) Patients who have undergone coronary artery bypass surgery in the last 3 months The study will be conducted with participants with chronic kidney disease diagnosed with coronary artery disease and dyslipidemia. Randomly selected participants of similar sizes will be randomly divided into 2 groups.

Group A (intervention group) will be asked to use 2 capsules containing 2000 mg (720 mg EPA, 480 mg DHA) omega 3 daily for 12 weeks. The total of these capsules taken in the morning and evening will provide the daily dose. Group B will be the control group. No supplements will be used in this group.

Anthropometric Measurements Individuals' body weight (kg), height (cm) measurements will be taken. Food Consumption Records Food consumption records will be taken from all individuals participating in the study at the beginning of the study in order to determine the daily energy and nutrients taken by the participants with their diet. They will also be evaluated with the food consumption frequency form.

The energy and nutrient contents of the consumed foods will be calculated using the "Nutrition Information System (BeBis)" program.

Subjective Global Assessment (SGD) Subjective Global Assessment (SGD) is frequently used in the evaluation of nutritional status in renal failure patients. It is considered an easily applicable and reliable method. All participants in our study will be evaluated with Subjective Global Assessment.

Biochemical Parameters Blood samples will be taken after 8 hours of fasting for the analysis of biochemical parameters. In the blood samples taken from the participants in the intervention and control groups at the beginning and end of the study; Total cholesterol (mg/dL), LDL-C (mg/dL), HDL-C (mg/dL), triglyceride (mg/dL), CRP (mg/L), fasting blood glucose (mg/dL), calcium (mg/dL), phosphorus (mg/dL), sodium (mg/dL) potassium (mg/dL), Creatine, Urea, Uric acid, Homocysteine Inflammatory Biomarkers: IL-6, TNF-a Oxidative Stress Biomarkers: Superoxide dismutase (SOD), Malondialdehyde (MDA) concentrations will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with dyslipidemia
* Patients diagnosed with type 2 diabetes
* Patients with a history of coronary artery disease
* Patients with a glomerular filtration rate of 20-60 ml/min
* Patients with stage 2-4 chronic kidney disease
* Patients with a body mass index (BMI) of 18-30 kg/m2
* Patients aged 45-80
* Patients with an LDL cholesterol level of >70 mg/dl despite taking statin medications at the same dose for at least 3 months

Exclusion Criteria:

* Those with active inflammatory diseases
* Those taking anti-inflammatory medications, those with chronic inflammation such as active hepatitis or human immunodeficiency virus (HIV)(+)
* Those with liver disease - elevated liver enzymes
* Those undergoing dialysis treatment
* Those planning a transplant
* Those using fish oil or other antioxidant medications within the last 3 months
* Those who are pregnant or breastfeeding
* Those with neurological or psychiatric disorders
* Individuals consuming more than one serving of fish per week
* Patients at high risk of bleeding (those using bivalirudin)
* Patients who have undergone coronary artery bypass surgery within the last 3 months

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Change in serum oxidative stress, inflammation, and lipid profile | Baseline and 12 weeks
  To evaluate changes in serum oxidative stress biomarkers (SOD (Superoxide Dismutase), MDA (Malondialdehyde), inflammation biomarkers (IL-6 (Interleukin-6), TNF-α (Tumor Necrosis Alpha), CRP (C-Reactive Protein) and lipid profile (LDL-C, HDL-C, Total cholesterol, Triglycerides) and homocysteine parameters between baseline and the end of the 12-week intervention.

SECONDARY OUTCOMES:
Weight change | Baseline and 12 weeks
  Participants' weights (kg) will be measured at the beginning of the study and at the end of 12 weeks.
Change in dietary intake | Baseline
  To determine participants' daily energy and nutrient intake, food consumption records will be collected from all participants at the beginning of the study. They will also be assessed using a food frequency form.
  The energy and nutrient contents of consumed foods will be calculated using the "Nutrition Information System (BeBis)" program.
Height | Baseline
  At the beginning of the study, participants' heights will be measured in 'cm'.

OTHER OUTCOMES:
Change in Subjective Global Assessment (SGA) score | Baseline and 12 week
  The Subjective Global Assessment (SGA) is a validated clinical tool used to assess nutritional status, particularly in patients with chronic kidney disease. It incorporates information from a patient interview and physical examination, including weight change, dietary intake, gastrointestinal symptoms, functional capacity, comorbidities, and physical signs of malnutrition (muscle wasting, subcutaneous fat loss, edema).
  In this study, the SGA will be performed at baseline and after 12 weeks of intervention by trained healthcare professionals. Scores range from:
  A: Well-nourished
  B: Mild to moderate malnutrition
  C: Severe malnutrition

CONTACTS AND LOCATIONS:
Overall Officials: EDA BALCI, lecturer, Principal Investigator — İstanbul Beykent University
Locations (1):
- Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)